CLINICAL TRIAL: NCT04628832
Title: Nudging Providers to Curtail Dangerous Opioid Prescribing: A Trial to Investigate Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Southern California (Other); Minnesota Management and Budget Agency (Unknown); Minnesota Board of Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAT2489
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Opioid Use
Keywords: opioids; prescribing; benzodiazepines; gabapentinoids; clinical guidelines; overprescribing; Benzodiazepine Use; Gabapentin Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PMP Use Mandate (Experimental)
  Interventions: Behavioral: PMP Use Mandate Letter
- Prescribing Information (Experimental)
  Interventions: Behavioral: Prescribing Information Letter
- Prescribing Information + PMP Use Mandate (Experimental)
  Interventions: Behavioral: Prescribing Information + PMP Use Mandate Letter
- Control / As-Usual (No Intervention)

INTERVENTIONS:
Behavioral: PMP Use Mandate Letter — A letter with reminders about the mandate to check the PMP when prescribing opioids.
  Arms: PMP Use Mandate
Behavioral: Prescribing Information Letter — A letter with information about the prescriber's patients who received co-prescriptions. The letters will provide clinical background on the harms of co-prescribing and encourage prescribers to avoid co-prescribing in the future.
  Arms: Prescribing Information
Behavioral: Prescribing Information + PMP Use Mandate Letter — A letter combining the content of the PMP Use Mandate Letter and the Prescribing Information Letter. This letter will remind prescribers about the PMP use mandate and provide information about the prescriber's patients who received co-prescriptions.
  Arms: Prescribing Information + PMP Use Mandate

SUMMARY:
Despite an enormous policy response, opioid prescribing remains well above historical levels and harms from opioids continue to mount. Nearly all states have Prescription Monitoring Programs (PMPs) to facilitate safer prescribing of opioids and other drugs, but research suggests these systems only deliver benefits when health care professionals are required to use them. Even with PMP mandates in place, providers may be unaware of the dangers of co-prescribing opioids with benzodiazepines or gabapentinoids, which include increased risk of overdose and death. Working with the Minnesota state government, the investigators will mail letters to guideline-discordant opioid prescribers that either highlight an upcoming legally mandated requirement to check the PMP before prescribing an opioid, inform and educate providers about patients filling concurrent prescriptions and the dangers of such co-prescribing, or both. Study participants will be randomized to receive no intervention or one of the three treatment letters. Using administrative data, the investigators will track effects of the letters on not only prescribing but also PMP usage and queries. Findings form the multiplicity of treatment messages and outcomes will shed light on the mechanisms driving overprescribing. Results will inform future work by state and local policymakers to make opioid prescribing safer.

ELIGIBILITY:
Inclusion Criteria:

* Wrote concurrent prescription for opioids and benzodiazepines OR opioids and gabapentinoids

Exclusion Criteria:

* Specialization in oncology or palliative medicine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12000 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Count of Patients with Co-Prescriptions | 60 days
  The number of patients with co-prescriptions from the prescriber in the 60 days after the letters are sent.
Rate of Prescribers Checking PMP | 60 days
  Indicator for whether the prescriber checks the PMP at least once in the 60 days after the letters are sent.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Sacarny, PhD, Principal Investigator — Columbia University; Mireille Jacobson, PhD, Principal Investigator — University of Southern California; David Powell, PhD, Principal Investigator — RAND
Locations (2):
- United States (2):
  - Minnesota Board of Pharmacy, Minneapolis, Minnesota
  - Minnesota Management and Budget Agency, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No